CLINICAL TRIAL: NCT02941211
Title: Effectiveness and Safety Evaluation of Aqueduct -100 Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqueduct Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AQD 01-14
Record Dates: First submitted 2016-08-30; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Cervix Uteri Dilation
Keywords: cervix; cervical dilation; balloon catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aqueduct 100 dilation (Experimental): Uterine cervix dilation through Aqueduct-100 device
  Interventions: Device: Aqueduct -100

INTERVENTIONS:
Device: Aqueduct -100

SUMMARY:
Evaluation of efficacy and safety of using Aqueduct -100 - Cervical Dilator Device

DETAILED DESCRIPTION:
There are predominantly two major dilatation techniques that are employed in dilating the cervix. The first technique uses expansible dry solid material, such as laminaria (seaweed) is inserted into the cervix in its dried stiff form. In the cervix it comes into contact with body fluids that cause the laminaria to swell and enlarge the cervical cavity. The second more widespread procedure, involves the use of series of solid, rod like instruments of graduated diameter used in serial fashion by the physician (Hegar dilators). The physician first inserts a rod like dilator and replaces it with the dilator of next higher diameter. This procedure continues until adequate dilatation occurs.

The Problem is that each of the above-mentioned methods has its shortcomings: the use of the laminaria method (rarely done) requires preliminary patient visit, for insertion of the laminaria rod and is extremely slow and typically involves often as much as 10-12 hours for a significant amount of dilatation to occur.

The use of rod-like instruments (Hegar) requires general or regional anesthesia, when local anesthetics are used, the patient nevertheless frequently experiences a great amount of discomfort from the procedure. The mechanical dilatation of the cervix demands a large amount of longitudinal force that may damage or even puncture the cervix and the uterus.

Aqueduct 100 is a catheter for use in dilating various body cavities and especially the human cervix. The device will enable continuous, fast and safe dilatation of the cervix to a pre-determined diameter as a pre-procedure to intrauterine surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, females, 18 years of age or older.
* Subjects undergoing any process that requires dilation (intrauterine procedures)
* Subjects willing to sign informed consent form.

Exclusion Criteria:

* Subjects younger than 18 years of age
* Subject with sex transmitted diseases, or with infectious diseases (HIV, HCV).
* Subjects unwilling to sign the informed consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with dilation of cervix to the diameter needed to perform the intrauterine procedure using Aqueduct-100 device. | Through study completion, approximately 6 months
  The primary outcome of this study is to determine the efficacy of the Aqueduct-100 device to dilate the uterine cervices to the desired diameter.

SECONDARY OUTCOMES:
Occurrence of Adverse Events | Through study completion, approximately 6 months
  Safety evaluation of using Aqueduct-100

OTHER OUTCOMES:
Time frame required to reach desired cervical dilation from start time (insertion of device) to completion of dilation (removal of catheter) | Through study completion, approximately 6 months
  Duration of the dilation procedure.
Measurement of physicians' overall satisfaction with the device through the use of a questionnaire | Through study completion, approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Javier Vico, MD, Principal Investigator — Hospital General Santa Maria del Puerto, Cádiz; Javier Pantoja, MD, Study Director — Hospital General Santa Maria del Puerto, Cádiz
Locations (1):
- Hospital General Santa Maria del Puerto, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
An article has been published in the digital edition of "Hysteroscopy Newsletter"

REFERENCES:
- [Background] Mazza E, Nava A, Bauer M, Winter R, Bajka M, Holzapfel GA. Mechanical properties of the human uterine cervix: an in vivo study. Med Image Anal. 2006 Apr;10(2):125-36. doi: 10.1016/j.media.2005.06.001. Epub 2005 Sep 6. PMID 16143559
- [Background] Buhimschi, C.; Buhimschi, I.; Malinow, A.; Saade, G.; Garfield, R.; Weiner, C., The Forces of Labour. Fetal and Maternal Medicine Review 2003, 14 (4), 273-307.
- [Background] Myers KM, Paskaleva AP, House M, Socrate S. Mechanical and biochemical properties of human cervical tissue. Acta Biomater. 2008 Jan;4(1):104-16. doi: 10.1016/j.actbio.2007.04.009. Epub 2007 Sep 27. PMID 17904431
- [Background] Kenyon NJ, Stevens JC, Stewart P, Black MM, Clifford A. A critical investigation of the measurement of the force required to dilate the human uterine cervix. Clin Phys Physiol Meas. 1988 May;9(2):155-61. doi: 10.1088/0143-0815/9/2/008. PMID 3391017
- [Background] S. Febvay, S. Socrate and M.D. House. Biomechanical modeling of cervical tissue. A quantitative investigation of cervical funneling. Proceedings of the ASME 2003 International Mechanical Engineering Congress and Exposition, Washington, D.C., November 2003
- [Background] Arsenijevic S, Vukcevic-Globarevic G, Volarevic V, Macuzic I, Todorovic P, Tanaskovic I, Mijailovic M, Raicevic S, Jeremic B. Continuous controllable balloon dilation: a novel approach for cervix dilation. Trials. 2012 Oct 22;13:196. doi: 10.1186/1745-6215-13-196. PMID 23088906
- [Background] Nicolaides KH, Welch CC, MacPherson MB, Johnson IR, Filshie GM. Lamicel: a new technique for cervical dilatation before first trimester abortion. Br J Obstet Gynaecol. 1983 May;90(5):475-9. doi: 10.1111/j.1471-0528.1983.tb08947.x. PMID 6849849
- See also: Aqueduct-100 functioning — https://www.youtube.com/watch?v=nJY3Y-hpdyw